CLINICAL TRIAL: NCT01483651
Title: The Hepatic Glucose Response to Glucagon at Varying Insulin Levels: Implications for Closed Loop Glycemic Control.
Brief Title: Physiologic Response to Glucagon at Varying Insulin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: kw02
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; glucagon; insulin; dideuterated glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Glucagon; Glucagon-Like Peptide 1; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low, Medium and High insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at lowest level with glucagon administration.
  Second study is regular insulin infused at medium level with glucagon adminstration.
  Third study is regular insulin infused at highest level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin
- Low, High and Medium insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at lowest level with glucagon administration.
  Second study is regular insulin infused at highest level with glucagon adminstration.
  Third study is regular insulin infused at medium level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin
- Medium, Low and High insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at medium level with glucagon administration.
  Second study is regular insulin infused at lowest level with glucagon adminstration.
  Third study is regular insulin infused at highest level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin
- Medium, High and Low insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at medium level with glucagon administration.
  Second study is regular insulin infused at highest level with glucagon adminstration.
  Third study is regular insulin infused at lowest level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin
- High, Low and Medium insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at highest level with glucagon administration.
  Second study is regular insulin infused at lowest level with glucagon adminstration.
  Third study is regular insulin infused at medium level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin
- High, Medium and Low insulin infusion (Experimental): All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at highest level with glucagon administration.
  Second study is regular insulin infused at medium level with glucagon adminstration.
  Third study is regular insulin infused at lowest level with glucagon administration.
  Interventions: Drug: Glucagon; Drug: Insulin

INTERVENTIONS:
Drug: Glucagon — The first dose of glucagon will be delivered approximately one hour after infusion of IV insulin has started. The subsequent three doses will be delivered every two hours. The dosage will depend on the IV insulin infusion (50 units regular insulin in 499.5 mL 0.9% saline): Study 1) insulin 0.01 units/kg/hour and glucagon doses (ug): 10,25,45,70; Study 2) insulin 0.02 units/kg/hr and glucagon doses (ug): 25,45,70,100; Study 3) insulin 0.04 units/kg/hr and glucagon doses (ug): 45,70,100,135; Study 4) insulin 0.08 units/kg/hr and glucagon doses (ug): 70,100,135,175. Insulin levels and glucagon doses will be randomized. Glucagon will be reconstituted with 10 mL of sterile water and administered subcutaneously.
  Other Names: GlucaGen
Drug: Insulin — Insulin was administered at a low, medium or high infusion rate. The intervention sequence was randomly pre-determined for all participants.
  Other Names: Regular insulin

SUMMARY:
The purpose of this research study is to test how different levels of insulin block the effect of glucagon. Insulin is a hormone that lowers blood glucose. Glucagon raises blood glucose. Both are natural hormones made by people without diabetes. Sensor-based blood glucose control studies have been done by our research group using glucagon in small doses to prevent hypoglycemia (low blood sugar). However, sometimes glucagon does not work to raise blood sugar. The investigators believe this is because of too much insulin in the body. This study will help determine how different levels of insulin in the body affect the ability of glucagon to raise blood sugar.

DETAILED DESCRIPTION:
We investigators have been working on the development of a closed loop (artificial endocrine pancreas) insulin and glucagon infusion system since 2005 and are part of the Juvenile Diabetes Research Foundation Artificial Pancreas Consortium. As part of our studies, we give small doses of glucagon to prevent hypoglycemia. As we assessed the success and failure of glucagon administration during these studies, we found the use of glucagon reduced the frequency of hypoglycemia by about 75%. However, the fact that approximately 25% of administrations of glucagon are ineffective remains a concern.

The primary question to be addressed by this study is, in the setting of low dose subcutaneous glucagon administration, how do plasma glucagon and plasma insulin quantitatively interact? In other words, as the rate of insulin administration is increased, how much more glucagon is necessary to overcome the effect of insulin to prevent hypoglycemia? This study is designed to address this question. Subjects will be brought in to a Legacy Hospital for four 10 hour experiments on each of four separate days. On each study day, there will be a continuous infusion of a different rate of IV Regular insulin in order to achieve different steady state free insulin levels. At each insulin level, there will be four subcutaneous glucagon doses given. Octreotide will be infused by IV at a constant rate to suppress endogenous production of glucagon. A stable glucose isotope will also be infused to allow for measurement of hepatic glucose production and glucose turnover. Arterialized venous blood glucose will be measured by the HemoCue Glucose 201 Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year
* Male or female subjects 21 to 65 years of age
* Current use of an insulin pump
* Willingness to sign informed consent and HIPAA documents and follow all study procedures

Exclusion Criteria:

* Pregnancy or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study
* Renal insufficiency (serum creatinine of 2.0 mg/dL or greater)
* Liver abnormalities: Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less than 3.3 g/dL; or serum bilirubin of over 2
* Adrenal insufficiency
* Hematocrit of less than or equal to 34%
* A history of cerebrovascular disease or coronary artery disease regardless of the time since occurrence
* Congestive heart failure, NYHA class III or IV
* Cardiac rhythm disturbance characterized by: 2nd or 3rd degree heart block, bradycardia of less than 50 bpm (exception of bradycardia in an aerobic athlete), tachycardia of greater than 100 bpm, or any arrhythmia judged by the investigator to be exclusionary
* Any active infection
* Active foot ulceration
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication
* Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator)
* Active malignancy, except basal cell or squamous cell skin cancers
* Major surgical operation within 30 days prior to screening
* Seizure disorder
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen
* Chronic usage of any immunosuppressive medication
* Current administration of oral or parenteral corticosteroids
* Use of an investigational drug within 30 days prior to screening
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000
* Allergy to glucagon
* Past history of pheochromocytoma or a family history of MEN 2, neurofibromatosis, or von Hippel-Lindau disease
* Insulin resistance requiring more than 200 units per day

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W Kenneth Ward, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Health System, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low, Medium and High Insulin Infusion Rate: All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at lowest level with glucagon administration.
  Second study is regular insulin infused at medium level with glucagon adminstration.
  Third study is regular insulin infused at highest level with glucagon administration.
- Low, High and Medium Insulin Infusion Rate: All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at lowest level with glucagon administration.
  Second study is regular insulin infused at highest level with glucagon adminstration.
  Third study is regular insulin infused at medium level with glucagon administration.
- Medium, Low and High Insulin Infusion Rate: All study subjects in this arm were randomized as follows:
  First study is regular insulin infused at medium level with glucagon administration.
  Second study is regular insulin infused at lowest level with glucagon adminstration.
  Third study is regular insulin infused at highest level with glucagon administration.
Period: Overall Study
Arm/Group | Low, Medium and High Insulin Infusion Rate | Low, High and Medium Insulin Infusion Rate | Medium, Low and High Insulin Infusion Rate | Medium, High and Low Insulin Infusion | High, Low and Medium Insulin Infusion | High, Medium and Low Insulin Infusion
Started | 1 | 3 | 2 | 1 | 2 | 2
Completed | 1 | 2 | 1 | 1 | 2 | 1
Not Completed | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Regular insulin given at each of three study visits with a different infusion rate at each visit, either low, medium or high insulin infusion with glucagon administration.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Glucose Above Baseline
Description: The change in the rate of glucose appearance will be assessed by measuring the stable glucose isotope (dideuterated glucose, D2) using a gas chromatography-mass spectrometry assay. The units of the area under the curve are defined as milligrams per kilogram of glucose, since the dependent variable is a rate of glucose production [mg/kg/min] measured over time [min]. The time variable therefore cancels out. Additionally, this area under the curve is being normalized per microgram of glucagon delivered.
Time Frame: 60 minutes after each glucagon administration
Measure: Mean (Standard Deviation); unit: mg/kg glucose per mcg glucagon
Groups:
- Low Insulin Infusion Rate: Regular insulin infused at lowest level of glucagon administration.
- Medium Insulin Infusion Rate: Regular insulin infused at medium level with glucagon administration.
- High Insulin Infusion Rate: Regular insulin infused at highest level with glucagon administration.
Arm/Group | Low Insulin Infusion Rate | Medium Insulin Infusion Rate | High Insulin Infusion Rate
Number analyzed (Participants) | 10 | 9 | 10
mg/kg glucose per mcg glucagon | 0.623 (0.3) | 0.59 (0.4) | 0.03 (0.16)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Low Insulin Infusion: Regular insulin infused at lowest level with glucagon administration.
- Medium Insulin Infusion: Regular insulin infused at medium level with glucagon administration.
- High Insulin Infusion: regular insulin infused at highest level with glucagon administration.
Arm/Group | Low Insulin Infusion | Medium Insulin Infusion | High Insulin Infusion
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 8/9 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Insulin Infusion (N=10) | Medium Insulin Infusion (N=9) | High Insulin Infusion (N=10)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 2 (3) | 3 (3)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
excessive thirst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
extravasation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
dermititis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ketosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes